CLINICAL TRIAL: NCT00895778
Title: Neuromuscular Blockade Improves Surgical Conditions
Acronym: NISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NISCO
Record Dates: First submitted 2009-04-29; First posted 2009-05-08 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular blockade; post-operative pain; post-operative pulmonary function
MeSH Terms: conditions — Pain, Postoperative | interventions — Neuromuscular Blockade; Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMB (Experimental): muscle relaxation (neuromuscular block) during laparoscopic cholecystectomy
  Interventions: Other: Neuromuscular blockade with rocuronium and reversal with sugammadex
- no NMB (Placebo Comparator): no muscle relaxation (neuromuscular block) during laparoscopic cholecystectomy
  Interventions: Other: Neuromuscular blockade with rocuronium and reversal with sugammadex

INTERVENTIONS:
Other: Neuromuscular blockade with rocuronium and reversal with sugammadex

SUMMARY:
This study is designed to test the clinical hypothesis that a neuromuscular block improves surgical conditions, operation time, and post-operative pain.

DETAILED DESCRIPTION:
Muscle relaxants are part of a balanced anesthesia regimen. So far, evidence is given that a neuromuscular block improves intubating conditions and protects against laryngeal morbidity. The doctrine, however, that a neuromuscular block improves surgical conditions and consequently patient care, is lacking any evidence based on clinical trials.

This study, therefore, is designed to test the clinically hypothesis that a neuromuscular block improves surgical conditions. One major problem in such a setting, however, is that it is difficult to measure what "good" or "better" surgical conditions are. We therefore suggest surrogates to test the hypothesis. The primary endpoint is the postoperative patient-controlled analgesic demand for adequate pain control. The secondary endpoints are the incidence of intraoperative events reflecting muscle relaxation during anesthesia, defined as movements of limbs or the abdominal wall, or as breathing, bucking or coughing against the ventilator, the incision-to-suture-time, the surgeon's and the anesthesiologist's opinion about the operating conditions assessed by a visual analogue scale (VAS), and the postoperative pulmonary function.

We will investigate patients scheduled for elective laparoscopic cholecystectomy under general anesthesia. The study is designed to allow optimal conditions to test the hypothesis. This results in two experimental groups representing two established anesthesia regimen (n = 25 per group). Patients of the group "no NMB" are anesthetized without any muscle relaxant. Patients of the group "NMB" are anesthetized using the same drugs as the "no NMB" group but additionally receive a neuromuscular blocking agent to induce a deep neuromuscular block from induction of anesthesia until skin suture.

Anesthesia will be induced with propofol and fentanyl. Airway will be managed using a ProSeal® Laryngeal mask which allows insertion of a gastric tube. Anesthesia will be maintained with desflurane inhalation and remifentanil infusion under BIS control. The group NMB will receive rocuronium to maintain a deep neuromuscular block (T2 < 2) until the fascia is sutured. Neuromuscular block will be reversed with sugammadex. Saline boli will be applied to the patients of the group "no NMB" every 25-35 min in order to keep the anesthesiologist blinded.

Post-operatively, in 15 min intervals during their stay and before discharge from the recovery room patients' level of consciousness will be assessed, and the updated Aldrete score will be obtained. In co-operative patients a 5-s head lift test, a 5-s arm lift test, swallowing of 20 ml water, and 5-s eye opening test will be performed. To achieve pain control, a microprocessor-controlled PCA system will be used.

The patients' respiratory function will be assessed before induction of anesthesia, 5 minutes after tracheal extubation, 30 minutes later in the postanesthesia care unit, and six hours later on the ward using a portable using spirometry device.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic cholecystectomy under general anesthesia
* Patients ASA physical status I - III
* Patients between 18 and 64 years
* Patients scheduled for general anesthesia with intubation using rocuronium
* Patients having given informed consent to the study

Exclusion Criteria:

* Anatomic and functional malformations with expected difficult intubation
* Known or suspected neuromuscular disease
* Significant hepatic or renal dysfunction
* Known or suspected history or family history of disposition to malignant hyperthermia
* Known or suspected allergy towards sugammadex, anesthetics, muscle relaxants, or other drugs used for general anesthesia
* Use of drugs that interfere with muscle relaxants
* Patients, included in another trial within the last 30 days
* Patients, with legal guidant
* Patients with contraindication towards the use of Sugammadex, neostigmine or glycopyrrolate
* Patients, which have already participated in a sugammadex trial
* Pregnant women (exclusion of pregnancy: postmenopausal status, negative beta-HCG screen, status post tubal ligation)
* Breastfeeding women
* Patients who are unable to understand or successfully administer a patient- controlled-analgesia (PCA) device

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postoperative patient-controlled analgesic demand for adequate pain control | Regular anesthesia time, approximately 1 hour

SECONDARY OUTCOMES:
Incidence of intraoperative muscle movements
Incision-to-suture-time
Surgeon's and anesthesiologist's opinion about the operating conditions assessed by a visual analogue scale (VAS)
Postoperative pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Blobner, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- [Background] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265
- [Derived] Blobner M, Frick CG, Stauble RB, Feussner H, Schaller SJ, Unterbuchner C, Lingg C, Geisler M, Fink H. Neuromuscular blockade improves surgical conditions (NISCO). Surg Endosc. 2015 Mar;29(3):627-36. doi: 10.1007/s00464-014-3711-7. Epub 2014 Aug 15. PMID 25125097